CLINICAL TRIAL: NCT05583851
Title: Digital Acceptance and Commitment Therapy (Digi-ACT): A Randomized Controlled Trial Pilot Assessing the Efficacy and Feasibility of Software-based Self-managed Intervention Targeting Subclinical Depression and Anxiety in Curative Cancer Patients Within Hong Kong
Brief Title: Investigating Whether Digital Acceptance Commitment Therapy Can Improve Mental Health for Hong Kong Cancer Patients Suffering From Depressive and Anxiety Symptoms.
Acronym: Digi-ACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hollo (Other)
Collaborators: OnCare Hong Kong (Unknown); The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Duncan Lim, Cognitive Scientist, Hollo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Project Axolotl
Record Dates: First submitted 2022-10-08; First posted 2022-10-18 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Depression, Anxiety; Quality of Life; Cancer
Keywords: Telemedicine; Acceptance and Commitment Therapy; Psycho-Oncology
MeSH Terms: conditions — Depression; Anxiety Disorders; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digi-ACT Intervention group (Experimental): 22 day long interactive mobile app intervention with daily activities. The intervention will include 5 total modules: psychoeducation on depression/anxiety and the cancer journey; acceptance; cognitive fusion; mindfulness; and committed valued living. There will be different games and reward components for the Through out the course of the intervention, participants will also do video journals to reflect on the different modules and activities they do.
  Interventions: Device: Acceptance and Commitment Therapy
- Psychoeducational Video Control group (Active Comparator): 22 day long mobile app where participants will be given a 15 minute long psychoeducational clip from a publicly available online seminar (from the Hong Kong College of Psychiatrists) on a bi-daily basis. Through out the course of the intervention, participants will also do video journals to reflect on the content of the different video clips.
  Interventions: Other: Psychoeducation Active Control

INTERVENTIONS:
Device: Acceptance and Commitment Therapy — Smartphone app guided and manualized version of acceptance and commitment therapy.
  Other Names: Digi-ACT; Digital Acceptance and Commitment Therapy
  Arms: Digi-ACT Intervention group
Other: Psychoeducation Active Control — Set of 11 public seminar videos regarding depression and anxiety. Each are 15 minutes long.
  Arms: Psychoeducational Video Control group

SUMMARY:
The goal of this clinical trial is to validate the use of digital Acceptance and Commitment Therapy (Digi-ACT) in Hong Kong curative cancer patients with depressive and anxiety symptoms. The main questions it aims to answer are:

* Can Digi-ACT reduce depressive or anxiety symptoms?
* Can Digi-ACT improved health-related quality of life?
* Is Digi-ACT an acceptable and feasible intervention for users?
* What are the factors that influence the success of Digi-ACT?
* Can the video journals used in Digi-ACT predict depressive symptoms?

Intervention group participants will install the Digi-ACT mobile application and undergo a 3-4 week long intervention. They will have to fill out questionnaires at baseline, immediately after the intervention, and at three month follow up to measure depression and anxiety symptoms, health-related quality of life, acceptability of the intervention, and other process outcomes related to the intervention itself.

Researchers will compare the outcomes with a group of participants that undergo a 3-4 week long period where they navigate a similar mobile platform that gives bi-daily psychoeducational videos that also fill out the same clinical questionnaires at baseline, post-intervention, and at three month follow up.

DETAILED DESCRIPTION:
Patients with cancer experience increased rates and severity of depression and anxiety symptoms. This could be due to difficulty dealing with the diagnostic process, treatment side effects, limited social opportunities, physical symptoms, and other cancer-related complications. Acceptance and Commitment Therapy (ACT) has proven to be effective in treating these symptoms for cancer patients. Compared to other evidence based therapies, such as second wave cognitive behavioral therapy (CBT), ACT has shown to have larger effect sizes and success in treating this population. One possible explanation could be due to the theoretical and practical approaches of ACT over traditional CBT. Traditional CBT aims to identify illogical thought patterns that are biased or distorted and try to change them, while ACT makes no attempt at changing these thought patterns and simply teaches the participant to accept and experience these thoughts, emotions, and sensations. For cancer patients, feelings of depression when faced with their own mortality, are unavoidable and could be invalidating if told they are "illogical" or "distorted". Therefore, ACT may have the advantage here in recognizing the severity of the cancer journey and providing an alternative way that does not try to change their experiences.

Furthermore, Hong Kong has a persisting mental health treatment gap due to insufficient mental health practitioners. Oftentimes, only moderate to severe cases of common mental disorders are addressed, thereby leaving milder cases untreated. A possible solution to such under-treatment is digital Health, which requires no additional practitioners and has shown promising results in past studies.

Therefore, we aim to test the efficacy, acceptability, and feasibility of a digitized version (mobile application) of ACT for cancer patients in Hong Kong.

We aim to answer several key questions with the current randomized controlled trial (RCT):

* Can Digi-ACT reduce depressive and anxiety symptoms from baseline to post-treatment and will this reduction be sustained at three month follow up?
* Can Digi-ACT improve health related quality of life from baseline to post-treatment and will this reduction be sustained at three month follow up?
* Is Digi-ACT perceived as an acceptable intervention prior to use? How about after use?
* Can different ACT process measures moderate the relationship between treatment and clinical outcomes?

Research assistants from Hollo will collaborate with Queen Mary Hospital's Oncological unit and Hong Kong Private Clinic: "Oncare" to recruit 50 Cancer patients for the pilot trial within the inclusion criteria. Participants will be screened at baseline for measures of depression and anxiety. Those that score mild or moderate will be invited to participate in the study. Upon providing informed consent, participants will be instructed to download the Hollo Digi-ACT mobile application.

Participants will be randomly allocated to either intervention or active control. Over 4 weeks, participants in the intervention group will be administered the digitized ACT on their mobile device while those in the active control will receive various educational mental health videos over the 4 weeks. After the completion of the intervention, participants will fill out the same clinical indexes and then a final time 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and above
* PHQ-9 score of 5 to 14
* BAI score of 8 to 25
* Fluent in Cantonese or Mandarin
* Diagnosed with stage 0 to 3 cancer
* Received surgery as primary treatment at least four months ago

Exclusion Criteria:

* Diagnosed with metastatic cancer (stage 4)
* Language/intellectual difficulties
* Prior diagnoses of other psychiatric conditions other than unipolar depression or anxiety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Depressive Symptoms severity as assessed by the 9 item Chinese Patient Health Questionnaire (PHQ-) from baseline to immediately after treatment and 3 month follow up | baseline, immediately after treatment, 3 month follow up
  The Chinese PHQ9 is a validated, self-report instrument that assesses depressive symptoms in the past 2 weeks. Possible scores range from 0 (no signs of depressive symptoms) to 27 (severe depressive symptoms).
Changes in Anxiety Symptoms severity as assessed by the Chinese Beck Anxiety Inventory (BAI) from baseline to immediately after treatment and 3 month follow up | baseline, immediately after treatment, 3 month follow up
  The 21 item Chinese (BAI) is a validated, self-report instrument that assesses anxiety symptoms in the past 2 weeks. Possible scores range from 0 (no signs of anxiety symptoms) to 63 (severe anxiety symptoms).
Changes in Quality of Life as assessed by the Chinese Functional Assessment of Cancer Therapy (FACT-G) from baseline to immediately after treatment and 3 month follow up | baseline, immediately after treatment, 3 month follow up
  The 27 item Chinese FACT-G is a validated, self-report instrument that assesses health related quality of life in the past week. Possible scores range from 0 (poor quality of life) to 108 (strong quality of life).

SECONDARY OUTCOMES:
Acceptability, measured by responses to 4 statements regarding expectations of the intervention at baseline and, immediately after treatment, and 3 month follow up. | baseline, immediately after treatment, 3 month follow up
  Acceptability, measured by responses to 4 statements regarding expectations of the intervention at baseline and, post-treatment, and 3 month follow up.
  The 4 item acceptability measure involve four statements that participants have to rate on a 1 (strongly agree) to 5 (strongly disagree). Statements presented at baseline are as follows:
  1. I expect to be satisfied with the content I received
  2. I expect the intervention facilitated emotional awareness
  3. I expect to learn something from the intervention
  4. I expect for what I learned to be relevant to my everyday life
  The four statements presented at post-treatment and 3 month follow up will be presented in past tense.
  Minimum score of 4 indicates strong acceptability and the maximum score of 20 indicates lack of acceptability.
Feasibility, measured by proportion of content completed by immediately after treatment | immediately after treatment
  For those in the intervention group, the digi-ACT content will include 5 modules. Therefore, feasibility for the intervention group will be calculated as the proportion of modules completed, with a score of 0 indicating no modules finished and a score of 1 indicating all modules completed. Similarly, for those in the control video group, there will be 11 videos and feasibility will be calculated as the proportion of these 11 videos viewed with the same minimum and maximum scores.

OTHER OUTCOMES:
Changes in Acceptance, as assessed by the Chinese White Bear Thought Suppression Inventory (WBSI) from baseline to immediately after treatment and 3 months follow up | baseline, immediately after treatment, 3 month follow up
  The 15 item Chinese WBSI measures the degree of thought suppression an individual presents. The inverse score from this measure could be interpreted as a measure of acceptance. Possible scores range from 15 (strong acceptance) to 75 (weak acceptance).
Changes in degree of Mindfulness as assessed by the Chinese Mindfulness Attention and Awareness Scale (CMAAS) from baseline to immediately after treatment and 3 month follow up | baseline, immediately after treatment, 3 month follow up
  The 15 item CMAAS is a validated, self-report instrument that assesses mindfulness. Total score is calculated as an average of the 15 items that are rated on a 1-6 likert scale. Therefore, the average minimum score starts at 1 (lower levels of mindfulness) and goes up to a maximum score of 6 (high levels of dispositional mindfulness.
Changes in cognitive fusion as assessed by the 9 item Chinese Cognitive Fusion Questionnaire (CFQ-9) from baseline to immediately after treatment and 3 month follow up | baseline, immediately after treatment, 3 month follow up
  The Chinese CFQ-9 is a validated, self-report instrument that assesses cognitive fusion. Possible scores range from 7 (low levels of cognitive fusion) to 63 (high levels of cognitive fusion)
Changes in valued living as assessed by the Chinese Valued Living Questionnaire (VLQ) from baseline to immediately after treatment and 3 month follow up | baseline, immediately after treatment, 3 month follow up
  The 10 item Chinese (VLQ) is a validated, self-report instrument that assesses the degree of valued living across 10 different domains. The maximum score of 100 indicates strong and alignment with values whereas a score of 0 would indicate weak alignment and weight placed on their 10 values.
Accuracy in video journal predicted PHQ-9 scores as assessed by an ai based video journal Within the baseline to immediately after treatment. | Between baseline and immediately after treatment
  A novel video journal measuring facial action units, pitch, and speech content will be used to predict a binary output on whether users present with depression or not. Participants, throughout the intervention or control video viewings, will have to shoot 2 minute videos to react and reflect on the contents of the intervention and videos.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Wing-lok Chan, MBBS, Principal Investigator — LKS Faculty of Medicine, HKU; Kevin Ka Ming Wong, MBBS, Principal Investigator — OnCare Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bai Z, Luo S, Zhang L, Wu S, Chi I. Acceptance and Commitment Therapy (ACT) to reduce depression: A systematic review and meta-analysis. J Affect Disord. 2020 Jan 1;260:728-737. doi: 10.1016/j.jad.2019.09.040. Epub 2019 Sep 10. PMID 31563072
- [Background] Barnes-Holmes Y, Hayes SC, Barnes-Holmes D, Roche B. Relational frame theory: a post-Skinnerian account of human language and cognition. Adv Child Dev Behav. 2001;28:101-38. doi: 10.1016/s0065-2407(02)80063-5. No abstract available. PMID 11605362
- [Background] Che, Lu, Chen, Chang. Validation of the Chinese Version of the Beck Anxiety Inventory. 台灣醫學. 1006; 447-454.
- [Background] Cheung G, Douwes G, Sundram F. Late-Life Suicide in Terminal Cancer: A Rational Act or Underdiagnosed Depression? J Pain Symptom Manage. 2017 Dec;54(6):835-842. doi: 10.1016/j.jpainsymman.2017.05.004. Epub 2017 Aug 12. PMID 28807701
- [Background] Cillessen L, Johannsen M, Speckens AEM, Zachariae R. Mindfulness-based interventions for psychological and physical health outcomes in cancer patients and survivors: A systematic review and meta-analysis of randomized controlled trials. Psychooncology. 2019 Dec;28(12):2257-2269. doi: 10.1002/pon.5214. Epub 2019 Sep 11. PMID 31464026
- [Background] Cotter DD. Psychometric evaluation of the Valued Living Questionnaire: Comparing distressed and normative samples. Western Michigan University. 2011.
- [Background] Deng Y, Li S, Tang, Zhu L, Ryan R, Brown K. Psychometric properties of the Chinese translation of the mindful attention awareness scale (MAAS). Mindfulness. 2012; 3(1), 10-14.
- [Background] Fitzpatrick KK, Darcy A, Vierhile M. Delivering Cognitive Behavior Therapy to Young Adults With Symptoms of Depression and Anxiety Using a Fully Automated Conversational Agent (Woebot): A Randomized Controlled Trial. JMIR Ment Health. 2017 Jun 6;4(2):e19. doi: 10.2196/mental.7785. PMID 28588005
- [Background] Gillanders DT, Bolderston H, Bond FW, Dempster M, Flaxman PE, Campbell L, Kerr S, Tansey L, Noel P, Ferenbach C, Masley S, Roach L, Lloyd J, May L, Clarke S, Remington B. The development and initial validation of the cognitive fusion questionnaire. Behav Ther. 2014 Jan;45(1):83-101. doi: 10.1016/j.beth.2013.09.001. Epub 2013 Sep 18. PMID 24411117
- [Background] Graham CD, Gouick J, Krahe C, Gillanders D. A systematic review of the use of Acceptance and Commitment Therapy (ACT) in chronic disease and long-term conditions. Clin Psychol Rev. 2016 Jun;46:46-58. doi: 10.1016/j.cpr.2016.04.009. Epub 2016 Apr 20. PMID 27176925
- [Background] Hayes SC. Buddhism and acceptance and commitment therapy. Cognitive and Behavioral Practice. 2002; 9(1), 58-66.
- [Background] Hayes SC. Get out of your mind and into your life: The new acceptance and commitment therapy. New Harbinger Publications. 2005.
- [Background] Hayes SC, Strosahl KD, Wilson KG. Acceptance and commitment therapy. Washington, DC: American Psychological Association. 2009.
- [Background] Hinz A, Krauss O, Hauss JP, Hockel M, Kortmann RD, Stolzenburg JU, Schwarz R. Anxiety and depression in cancer patients compared with the general population. Eur J Cancer Care (Engl). 2010 Jul;19(4):522-9. doi: 10.1111/j.1365-2354.2009.01088.x. Epub 2009 Dec 17. PMID 20030697
- [Background] Kim J, Shin W. How to do random allocation (randomization). Clin Orthop Surg. 2014 Mar;6(1):103-9. doi: 10.4055/cios.2014.6.1.103. Epub 2014 Feb 14. PMID 24605197
- [Background] Kioskli K, Scott W, Winkley K, Godfrey E, McCracken LM. Online Acceptance and Commitment Therapy for People with Painful Diabetic Neuropathy in the United Kingdom: A Single-Arm Feasibility Trial. Pain Med. 2020 Nov 1;21(11):2777-2788. doi: 10.1093/pm/pnaa110. PMID 32358608
- [Background] Li H, Wong CL, Jin X, Chen J, Chong YY, Bai Y. Effects of Acceptance and Commitment Therapy on health-related outcomes for patients with advanced cancer: A systematic review. Int J Nurs Stud. 2021 Mar;115:103876. doi: 10.1016/j.ijnurstu.2021.103876. Epub 2021 Jan 12. PMID 33517079
- [Background] Lin J, Paganini S, Sander L, Luking M, Ebert DD, Buhrman M, Andersson G, Baumeister H. An Internet-Based Intervention for Chronic Pain. Dtsch Arztebl Int. 2017 Oct 13;114(41):681-688. doi: 10.3238/arztebl.2017.0681. PMID 29082858
- [Background] Luoma JB, Hayes SC, Walser RD. Learning ACT: An acceptance & commitment therapy skills-training manual for therapists. New Harbinger Publications. 2007.
- [Background] Masuda A, Hayes SC, Sackett CF, Twohig MP. Cognitive defusion and self-relevant negative thoughts: examining the impact of a ninety year old technique. Behav Res Ther. 2004 Apr;42(4):477-85. doi: 10.1016/j.brat.2003.10.008. PMID 14998740
- [Background] Men VY, Emery CR, Yip PSF. Characteristics of cancer patients who died by suicide: A quantitative study of 15-year coronial records. Psychooncology. 2021 Jul;30(7):1051-1058. doi: 10.1002/pon.5634. Epub 2021 Mar 2. PMID 33655563
- [Background] Menin J, de Blasio B. New York city mobile services study. Research Brief, Department of Consumer Affairs, New York City. 2015.
- [Background] Ost LG. The efficacy of Acceptance and Commitment Therapy: an updated systematic review and meta-analysis. Behav Res Ther. 2014 Oct;61:105-21. doi: 10.1016/j.brat.2014.07.018. Epub 2014 Aug 19. PMID 25193001
- [Background] Pitman A, Suleman S, Hyde N, Hodgkiss A. Depression and anxiety in patients with cancer. BMJ. 2018 Apr 25;361:k1415. doi: 10.1136/bmj.k1415. No abstract available. PMID 29695476
- [Background] Rodriguez MA, Jia K, Qian MY. White Bear Suppression Inventory: Structure, reliability and validity of the Chinese version. Chinese Journal of Clinical Psychology. 2012.
- [Background] Razzouk R, Shute V. What is design thinking and why is it important?. Review of educational research. 2012; 82(3): 330-348.
- [Background] Simister HD, Tkachuk GA, Shay BL, Vincent N, Pear JJ, Skrabek RQ. Randomized Controlled Trial of Online Acceptance and Commitment Therapy for Fibromyalgia. J Pain. 2018 Jul;19(7):741-753. doi: 10.1016/j.jpain.2018.02.004. Epub 2018 Mar 2. PMID 29481976
- [Background] Tatrow K, Montgomery GH. Cognitive behavioral therapy techniques for distress and pain in breast cancer patients: a meta-analysis. J Behav Med. 2006 Feb;29(1):17-27. doi: 10.1007/s10865-005-9036-1. Epub 2006 Jan 7. PMID 16400532
- [Background] Trompetter HR, Bohlmeijer ET, Veehof MM, Schreurs KM. Internet-based guided self-help intervention for chronic pain based on Acceptance and Commitment Therapy: a randomized controlled trial. J Behav Med. 2015 Feb;38(1):66-80. doi: 10.1007/s10865-014-9579-0. Epub 2014 Jun 13. PMID 24923259
- [Background] van de Graaf DL, Trompetter HR, Smeets T, Mols F. Online Acceptance and Commitment Therapy (ACT) interventions for chronic pain: A systematic literature review. Internet Interv. 2021 Oct 1;26:100465. doi: 10.1016/j.invent.2021.100465. eCollection 2021 Dec. PMID 34660209
- [Background] Wang W, Bian Q, Zhao Y, Li X, Wang W, Du J, Zhang G, Zhou Q, Zhao M. Reliability and validity of the Chinese version of the Patient Health Questionnaire (PHQ-9) in the general population. Gen Hosp Psychiatry. 2014 Sep-Oct;36(5):539-44. doi: 10.1016/j.genhosppsych.2014.05.021. Epub 2014 Jun 6. PMID 25023953
- [Background] Wegner DM, Zanakos S. Chronic thought suppression. J Pers. 1994 Dec;62(4):616-40. doi: 10.1111/j.1467-6494.1994.tb00311.x. PMID 7861307
- [Background] Wei-Chen Z, Yang J, Li X, Hui-Na G, Zhuo-Hong Z. Reliability and validity of the Chinese version of the Cognitive Fusion Questionnaire. Chinese Mental Health Journal. 2014;28(1): 40-44.
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Background] Yu CL, Fielding R, Chan CL, Tse VK, Choi PH, Lau WH, Choy DT, O SK, Lee AW, Sham JS. Measuring quality of life of Chinese cancer patients: A validation of the Chinese version of the Functional Assessment of Cancer Therapy-General (FACT-G) scale. Cancer. 2000 Apr 1;88(7):1715-27. PMID 10738232
- [Background] Yu X, Tam WW, Wong PT, Lam TH, Stewart SM. The Patient Health Questionnaire-9 for measuring depressive symptoms among the general population in Hong Kong. Compr Psychiatry. 2012 Jan;53(1):95-102. doi: 10.1016/j.comppsych.2010.11.002. Epub 2010 Dec 28. PMID 21193179
- [Background] Zhao C, Lai L, Zhang L, Cai Z, Ren Z, Shi C, Luo W, Yan Y. The effects of acceptance and commitment therapy on the psychological and physical outcomes among cancer patients: A meta-analysis with trial sequential analysis. J Psychosom Res. 2021 Jan;140:110304. doi: 10.1016/j.jpsychores.2020.110304. Epub 2020 Nov 20. PMID 33248396